CLINICAL TRIAL: NCT07273877
Title: Main Objective: To Evaluate the Long-term Safety and Efficacy of Using the Netrod-RDN Renal Artery Radiofrequency Ablation System in Treating Patients With Refractory Hypertension and Those With Hypertension Who Are Intolerant to Medication in the Real-world Setting
Brief Title: A Real-World Study on the Treatment of Hypertension With Netrod-RDN Renal Artery Radiofrequency Ablation System
Status: Enrolling by invitation | Type: Observational
Sponsor: Shanghai Golden Leaf MedTec Co. Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: MLWY-S240801
Record Dates: First submitted 2025-06-23; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Refractory hypertension and hypertension with drug intolerance Patient: For patients who have been taking more than three types of antihypertensive drugs (including one diuretic) for more than 3 months and whose blood pressure has not been controlled adequately; drug intolerance refers to patients who cannot tolerate the medication due to drug contraindications or adverse drug reactions.
  Interventions: Device: Percutaneous nephrolysis combined with sympathetic nerve ablation (RDN) procedure

INTERVENTIONS:
Device: Percutaneous nephrolysis combined with sympathetic nerve ablation (RDN) procedure — The disposable mesh renal artery radiofrequency ablation catheter is a spiral-arranged 6-point mesh system. Once The use of a meshed renal artery radiofrequency ablation catheter in combination with a dedicated renal artery radiofrequency ablation device delivers radiofrequency energy to the inner wall of the renal artery, generating appropriate high temperatures to damage or partially damage the renal sympathetic nerves. This device has real-time temperature, power and impedance monitoring functions, providing real-time ablation feedback. It also has the function of real-time recording of ablation data and saving the data.

SUMMARY:
This study is an observational one, collecting real-world data generated in routine clinical treatment. The Netrod-RDN renal artery radiofrequency ablation system (including the renal artery radiofrequency ablation device and the disposable mesh renal artery radiofrequency ablation catheter) produced and provided by Shanghai Meiliweiye Medical Technology Co., Ltd. was used to perform percutaneous renal denervation (RDN) on patients with refractory hypertension and drug intolerance in the real world. Refractory hypertension is defined as patients whose blood pressure remains uncontrolled despite taking three or more antihypertensive drugs (including one diuretic) for more than three months; drug intolerance refers to patients who have contraindications to drugs or cannot tolerate drug administration due to adverse drug reactions.

DETAILED DESCRIPTION:
All the subjects who were enrolled and received RDN treatment were followed up until 36 months after the surgery. Blood pressure was measured and the antihypertensive effect was evaluated at regular intervals at 7 days after RDN or before discharge (whichever came first), 30 days (±7 days) after the surgery, 3 months (±14 days), 6 months (±30 days), 12 months (±30 days), 24 months (±30 days), and 36 months (±30 days) during the follow-up. Dynamic safety data monitoring was conducted for the subjects throughout the entire study process.

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients who have already used or are planning to use the Netrod-RDN renal artery radiofrequency ablation system for RDN surgery;
* (2) Patients understand the requirements and treatment of this clinical study, agree to follow the requirements of this clinical study for follow-up, and sign the informed consent form before undergoing any special examinations and operations related to the study.

Exclusion Criteria:

* Patients with contraindications for RDN surgery and/or those who the researchers consider unsuitable for RDN or who do not wish to participate in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with refractory hypertension and those with drug intolerance in the real world
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in 24-hour Ambulatory Blood Pressure (including both systolic and diastolic BP) | Time Frame: Baseline to Month 6 post-procedure.

SECONDARY OUTCOMES:
Change from Baseline in Office Blood Pressure (including both systolic and diastolic BP) | Baseline to Day 7 or hospital discharge (whichever occurs first), and Months 1, 3, 6, 12, 24, and 36 post-procedure.
Change from Baseline in 24-hour Ambulatory Blood Pressure (including both systolic and diastolic BP) | Baseline to 3, 12, 24, and 36 months post-procedure
Change from Baseline in Home Blood Pressure (including both systolic and diastolic BP) | Time Frame: Baseline to Months 1, 3, 6, 12, 24, and 36 post-procedure.
Change from Baseline in Antihypertensive Medication Load (calculated based on the dosage and types of antihypertensive agents). | Baseline to Day 7 or hospital discharge (whichever occurs first), and Months 1, 3, 6, 12, 24, and 36 post-procedure.
Proportion of Participants Achieving Blood Pressure Targets (Office, Home, and 24-hour Ambulatory; including both systolic and diastolic BP) | At the same assessment time points as the above BP measurements (office, home, and 24-hour ambulatory BP).
  Office BP target <140/90 mmHg or <130/80 mmHg; Home BP target <135/85 mmHg; 24-hour ambulatory BP target <130/80 mmHg.
24-hour Time in Target Range for Ambulatory Blood Pressure (percentage of time meeting daytime <135/85 mmHg and nighttime <120/70 mmHg thresholds) | Months 6, 12, and 36 post-procedure.
Change from Baseline in SF-12 Health-Related Quality of Life Score (for heart failure subgroup only) | Baseline to Months 12 and 36 post-procedure.
  The SF-12 Health-Related Quality of Life Score includes Physical Component Summary (PCS) and Mental Component Summary (MCS) scores, using a norm-based system and not bonded by an absolute maximum or minimum, a higher SF-12 score on either the PCS or the MCS means a better health-related quality of life. Comparing the SF-12 scores before and after treatment can evaluate the improvement of the treatment on patient's daily quality of life.
Change from Baseline in Six-Minute Walk Distance (meters; heart failure subgroup only) | Baseline to Months 6, 12, 24, and 36 post-procedure.
Periprocedural major adverse event (MAE) rate | Baseline to 30 days post-procedure
  All-cause death;
  ESRD (eGFR <15 mL/min/1.73 m² or initiation of dialysis) or CKD progression (>50% decrease in eGFR or >50% increase in serum creatinine from baseline);
  Major thromboembolic events causing end-organ damage or requiring intervention to prevent it;
  Major vascular complications requiring surgical or endovascular intervention, including renal artery perforation, dissection, aneurysm, etc., and access-site vascular complications requiring intervention (e.g., hematoma, bleeding, arteriovenous fistula, etc.);
  Hospitalization for hypertensive crisis or significant hypotension not attributable to poor adherence to antihypertensive therapy;
  New renal artery stenosis >70% (confirmed by angiography).
Safety event rates | Baseline to Month 36 post-procedure
  All-cause mortality;
  ESRD (CKD stage 5; eGFR <15 mL/min/1.73 m²) or CKD progression (>50% decrease in eGFR from baseline or >50% increase in serum creatinine from baseline);
  Major thromboembolic events causing end-organ damage or requiring intervention to prevent it;
  Hospitalization for hypertensive crisis or clinically significant hypotension (not attributable to poor adherence to antihypertensives);
  New renal artery stenosis >70% (confirmed by angiography);
  New-onset acute coronary syndrome (ACS);
  New stroke, transient ischemic attack (TIA), or other major cerebrovascular events;
  Rehospitalization for worsening heart failure (HF subgroup only).

CONTACTS AND LOCATIONS:
Locations (1):
- Capital Medical University Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No